CLINICAL TRIAL: NCT06931652
Title: A Phase 2 Study Evaluating Epcoritamab in Subjects With Relapsed and Refractory Primary Diffuse Large B-cell Lymphoma of the CNS Treated With Lenalidomide and Rituximab
Brief Title: Study of Epcoritamab in R/R Primary Diffuse Large B-cell Lymphoma of the CNS Treated With Lenalidomide and Rituximab
Acronym: E-REVRI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-REVRI
Record Dates: First submitted 2025-04-07; First posted 2025-04-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Primary CNS Lymphoma (PCNSL)
Keywords: primary CNS lymphoma; treatment for primary CNS lymphoma; epcoritamab treatment; rituximab and lenalidomide treatment; Primary CNS Lymphoma (PCNSL)

STUDY DESIGN:
Intervention Model Description: This open-label, multicenter, single-arm phase II study is designed to assess the efficacy / safety of sub-cutaneous epcoritamab in subjects with relapsed or refractory diffuse large B-cell primary CNS Lymphoma (principal cohort: PCNSL) and relapsed or refractory primary vitreo-retinal lymphoma (exploratory cohort: PVRL) treated with oral lenalidomide and intravenous rituximab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental/epcoritamab (Experimental): Investigational Medicinal Product (IMP): Epcoritamab will be used during induction phase and Maintenance phase.
  Auxiliary Medicinal Products (AMP): Rituximab and Lenalidomide
  Standard use for AMP is:
  Induction:
  At cycle 1: Rituximab IV 375mg/m2 Day 1, 8, 15, 22; Lenalidomide 20mg oral route Day 1-Day 21 At cycle 2-3: Day 1: rituximab IV 375mg/m2; Lenalidomide 20mg oral route Day 1-Day 21 At cycle 4-8: Day 1: rituximab IV 375mg/m2; Lenalidomide 20mg oral route Day 1-Day 21
  Maintenance:
  At cycle 9-20: Day 1: Lenalidomide 20mg oral route Day 1-D21 (12 cycles corresponding to one year of maintenance treatment)
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Epcoritamab Investigational Medicinal Product (IMP): Epcoritamab will be used during induction phase and Maintenance phase.

SUMMARY:
The purpose of this phase 2 study is to evaluate the efficacy and safety of epcoritamab in subjects with relapsed or refractory primary diffuse large B-cell lymphoma of the Central Nervous System treated with rituximab and lenalidomide.

DETAILED DESCRIPTION:
Primary CNS DLBCL has an altered prognostic compared to systemic DLBCL mostly due to an increased relapse rate. PCNSL patients for whom the global prognostic remains poor, calling for improved treatment at relapse.

Considering the good results of R2 regimen in R/R PCNSL and the efficacy and favorable safety profile of epcoritamab in R/R systemic DLBCL, the addition of Epcoritamab to the combination of R2 might significantly improve the prognosis of PCNSL patients at relapse. In addition, it is expected that IMiDs could potentially increase the efficiency of epcoritamab by stimulating the immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or their legally acceptable representative/trusted person) who understand and voluntarily signs and dates an informed consent form prior to any study-specific assessments/procedures being conducted.
2. Subject ≥ 18 years old at the time of signing the informed consent form (ICF)
3. Confirmed histology of primary diffuse large B-cell lymphoma of the CNS (according to the 2022 WHO classification) or confirmed cytology of primary vitreoretinal diffuse large B-cell lymphoma, with CD20 positivity in immunohistochemical staining or flow cytometry at any point in the disease history.
4. Subjects with relapsed or refractory (R/R) PCNSL or PVRL after at least one line of systemic therapy. Subject with R/R PCNSL must have previously received at least high dose methotrexate. Subject with R/R PVRL must have received either intravenous high dose methotrexate or intraocular methotrexate (PVRL cohort). Subjects can have received radiotherapy or intensive chemotherapy with hematopoietic stem cell rescue as part of treatment of the PCNSL or PVRL.
5. ECOG performance status 0 to 2.
6. Estimated minimum life expectancy of ≥ 2 months.
7. R/R PCNSL subjects with evaluable disease on brain MRI.
8. Able to swallow capsules (stomach tube not allowed)
9. Adequate hematopoietic function:

   * Absolute neutrophil count of ≥ 1.0 G/L without G-CSF support for at least 7 days before screening
   * Platelet count of ≥ 50 G/L without platelet transfusion within 7 days before screening
   * Hemoglobin ≥ 8.0 g/dL without RBC transfusion within 7 days before screening
10. Adequate renal function: calculated by Cockcroft-Gault equation creatinine clearance > 40 ml/min. Subjects with calculated creatinine clearance > 40 and < 60ml/min lenalidomide dose will be adjusted.
11. Adequate liver function: Serum total bilirubin level ≤ 2.0 mg/dl [34 µmol/L] (unless bilirubin rise is due to Gilbert's syndrome) and serum transaminases (AST or ALT) ≤ 3 upper normal limits.
12. Able to understand teratogenic risks of the treatment (Lenalidomide).
13. Women of childbearing potential (WOCBP) should agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study treatment, 2) while participating in the study, 3) dose interruptions, and 4) for at least 12 months after the final dose of rituximab, or for at least 12 months after the final dose of epcoritamab, or for at least 28 days after the final dose of lenalidomide . WOCBP should also agree to abstain from breastfeeding during study participation and for at least 4 months after discontinuation of all study treatments.
14. WOCBP should have a negative serum (beta-hCG) pregnancy test at screening and a negative serum or urine pregnancy test before treatment administration on Day 1 of every cycle.
15. Women should agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire study, until 12 months after the last administration of study treatment.
16. Man who is sexually active with a female of reproductive potential and has not had a vasectomy should agree to use a highly effective / an acceptable method of birth control (ie, condom) and must agree not to donate sperm, until 28 days after the final dose of lenalidomide and/or until 12 months after the final dose of epcoritamab and rituximab.
17. Subject covered by any social security system (France).
18. Subject (or their legally acceptable representative/trusted person) who understands and speaks one of the country official languages unless local regulation authorizes independent translators.

Exclusion criteria:

Subject who meets any of the following criteria should be excluded from enrollment in the study:

1. T-cell lymphoma.
2. Cerebral localization of a systemic lymphoma.
3. Prior history of organ transplantation or other cause of severe immunodeficiency.
4. Known Human Immunodeficiency Virus (HIV) or Positive HTLV1 serology.
5. Active Hepatitis B Virus (HBV) infection (DNA PCR-positive) or active hepatitis C Virus (HCV) infection (RNA PCR-positive). Subjects with evidence of prior HBV infection but who are PCR-negative are permitted in the study but should receive prophylactic antiviral therapy. Subjects who received treatment for HCV infection that was intended to eradicate the virus may participate if hepatitis C RNA levels are undetectable.
6. Persistent SARS-CoV-2 infection. Subjects who have had or currently have a SARS-CoV-2 infection must demonstrate symptom resolution and provide a negative nasopharyngeal PCR test at time of inclusion. Both of these requirements must be met for the subject to be considered clear of the virus.
7. Impossibility to follow the calendar of exams because of geographic, social, or psychological reasons.
8. Active malignancy other than the one treated in this Study. Prior history of malignancies (other than inclusion diagnosis) unless the subject has been free of the disease for ≥ 2 years. However, subjects with the following history/concurrent conditions are allowed:

   1. Non-invasive basal cell or epidermoid carcinoma
   2. In situ Carcinoma of the cervix
   3. In situ Carcinoma of the breast
   4. Non-invasive, superficial bladder cancer
   5. Incidental histologic finding of prostate cancer (T1a or T1b) using the tumor, nodes, metastasis [TNM] clinical staging system
   6. Any curable cancer with a complete response of >2 years duration
9. Known or suspected hypersensitivity to the active substance or to any of the excipients.
10. Any previous treatment with CAR-T therapy within 30 days prior to enrollment.
11. Receiving immunosuppressive therapy, including more than the equivalent of 20 mg of prednisolone daily, unless for control of lymphoma or intermittent prophylaxis/treatment of allergic reactions.
12. Any previous treatment with a bispecific antibody targeting CD3 and CD20 and/or with lenalidomide, regardless of the time and duration.
13. Seizure disorder requiring anti-epileptic therapy unless related to lymphoma.
14. Vaccination with live, attenuated vaccines within 28 days prior of enrollment (except severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine). Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Experimental and/or non-authorized SARS-CoV-2 vaccinations are not allowed.
15. Use of any standard or experimental anti-cancer drug therapy within 28 days of the start (Day 1) of study treatment.
16. Major surgery within 4 weeks prior to enrollment
17. Clinically significant cardiovascular disease, including:

    1. Myocardial infarction within 1 year prior to enrollment, or unstable or uncontrol disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV) cardiac arrhythmia (CTCAE Version 5.0 Grade 2 or higher), or clinically significant ECG abnormalities.
    2. Stroke within 6 months prior to enrollment.
18. Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
19. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring systemic treatment at time of enrollment.
20. Contraindication to all uric acid lowering agents.
21. Clinically significant liver disease, including active hepatitis, current alcohol abuse, or cirrhosis.
22. Active tuberculosis or history of treatment for active tuberculosis within the past 12 months.
23. Receiving immunostimulatory agent.
24. Prior allogeneic hematopoietic stem cell transplantation.
25. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with participation in this clinical study (according to the investigator's decision).
26. Subject deprived of his/her liberty by a judicial or administrative decision.
27. Subject hospitalized without consent.
28. Adult subject under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The best Objective Response rate (ORR) in the R/R PCNSL cohort | after 8 months or before in case of permanent treatment discontinuation
  Objective Response rate

SECONDARY OUTCOMES:
Objective response rate (CR + CRu + PR) | after 8 months or before in case of permanent treatment discontinuation
  Objective response rate
Best objective response rate (CR + CRu + PR) in the PVRL cohort | after 8 months or before in case of permanent treatment discontinuation
  Objective response rate
Objective response rate (CR + CRu + PR) in the PVRL cohort | after 8 months or before in case of permanent treatment discontinuation
  Objective response rate
Best complete response rate (CR+CRu) | after 8 months or before in case of permanent treatment discontinuation
  Best complete response rate
Time to objective response (TTR) according to IPCG recommendations | 44 months after first patient in
  Time to objective response
Progression-free survival (PFS) according to IPCG recommendations | 56 months after first patient in
  Progression-free survival
Duration of response (DOR) according to IPCG recommendations | 56 months after first patient in
  Duration of response
Overall Survival (OS) | 56 months after first patient in
  Overall Survival
Time to next treatment (TTNT) | 56 months after first patient in
  Time to next treatment
Incidence and severity of AEs, special focus on ICANS, CRS and TLS | 56 months after first patient in
  Incidence and severity
Incidence and severity of changes in laboratory values | 44 months after first patient in
  Incidence and severity
Incidence of dose delay and treatment discontinuation | 44 months after first patient in
  Incidence of dose delay
Time to deterioration in physical functioning - EORTC QLQ-C30 | 44 months after First Patient In
  EORTC QLQ-C30 quality of life questionnaire. 30 questions using a scale of 4: from 1 (not at all) to 4 (very much). (lower score (worse): 120 and higher score (better): 30)
Cognitive evaluation with MoCA test | 56 months after first patient in
  10 questions / topics with different scores (between 1 and 6) and with a total score /30" (lower score (worse): 0 and higher score (better)
Time to deterioration in physical functioning - QLQ-HG29 | 44 months after First Patient In
  QLQ-HG29 Questionnary of Life: 29 additional questions using a scale of 4: from 1 (not at all) to 4 (very much). (lower score (worse): 116 and higher score (better): 29)
Cognitive evaluation with with BEARNI test | 56 months after first patient in
  5 questions / topics with different scores (between 5 and 8) and with a total score /30" (lower score (worse): 0 and higher score (better): 30)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Pr. Ghesquieres, MD, Principal Investigator — HCL - Hôpital Lyon Sud - Service d'Hématologie - 165 Chemin du Grand Revoyet, 69310 Pierre-Bénite - France; Gabriel Dr. Antherieu, MD, Principal Investigator — HCL - Hôpital Lyon Sud - Service d'Hématologie - 165 Chemin du Grand Revoyet, 69310 Pierre-Bénite - France
Locations (13):
- France (13):
  - INSTITUT BERGONIE - Service d'Oncologie Médicale, Bordeaux
  - INSTITUT D'HEMATOLOGIE DE BASSE NORMANDIE - Service Hématologie, Caen
  - CHU ESTAING - Service Thérapie Cellulaire et Hématologie Clinique, Clermont-Ferrand
  - CHU DE LILLE - HOPITAL CLAUDE HURIEZ - Service des Maladies du Sang, Lille
  - CHR DE MARSEILLE - CHU TIMONE - Service de Neuro-Oncologie, Marseille
  - CHRU DE NANCY - HOPITAL CENTRAL - Service de Neurologie, Nancy
  - GHU PITIE-SALPETRIERE - CHARLES FOIX - Service Neurologie, Paris
  - HOPITAL DE LA PITIE SALPETRIERE - Service Hématologie Clinique, Paris
  - CHU LYON-SUD - Hématologie Clinique, Pierre-Bénite
  - CHU PONTCHAILLOU - Hématologie Clinique, Rennes
  - INSTITUT CURIE - SITE SAINT-CLOUD - Service Hématologie, Saint-Cloud
  - IUCT ONCOPOLE - Service Hématologie, Toulouse
  - CHU BRETONNEAU - Service Cancérologie - Hématologie et Thérapie Cellulaire, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghesquieres H, Chevrier M, Laadhari M, Chinot O, Choquet S, Molucon-Chabrot C, Beauchesne P, Gressin R, Morschhauser F, Schmitt A, Gyan E, Hoang-Xuan K, Nicolas-Virelizier E, Cassoux N, Touitou V, Le Garff-Tavernier M, Savignoni A, Turbiez I, Soumelis V, Houillier C, Soussain C. Lenalidomide in combination with intravenous rituximab (REVRI) in relapsed/refractory primary CNS lymphoma or primary intraocular lymphoma: a multicenter prospective 'proof of concept' phase II study of the French Oculo-Cerebral lymphoma (LOC) Network and the Lymphoma Study Association (LYSA)dagger. Ann Oncol. 2019 Apr 1;30(4):621-628. doi: 10.1093/annonc/mdz032. PMID 30698644
- [Result] Top FU, Usta T, Gucesan S. [Determining headache characteristics among Health Sciences Faculty students and evaluating the cultural beliefs affecting their treatment selection(s)]. Agri. 2010 Jan;22(1):13-20. Turkish. PMID 20209410
- [Result] Houillier C, Dureau S, Taillandier L, Houot R, Chinot O, Molucon-Chabrot C, Schmitt A, Gressin R, Choquet S, Damaj G, Peyrade F, Abraham J, Delwail V, Gyan E, Sanhes L, Cornillon J, Garidi R, Delmer A, Al Jijakli A, Morel P, Waultier A, Paillassa J, Chauchet A, Gastinne T, Laadhari M, Plissonnier AS, Feuvret L, Cassoux N, Touitou V, Ricard D, Hoang-Xuan K, Soussain C; LOC Network for CNS Lymphoma. Radiotherapy or Autologous Stem-Cell Transplantation for Primary CNS Lymphoma in Patients Age 60 Years and Younger: Long-Term Results of the Randomized Phase II PRECIS Study. J Clin Oncol. 2022 Nov 10;40(32):3692-3698. doi: 10.1200/JCO.22.00491. Epub 2022 Jul 14. PMID 35834762
- [Result] O'Neill BP, Decker PA, Tieu C, Cerhan JR. The changing incidence of primary central nervous system lymphoma is driven primarily by the changing incidence in young and middle-aged men and differs from time trends in systemic diffuse large B-cell non-Hodgkin's lymphoma. Am J Hematol. 2013 Dec;88(12):997-1000. doi: 10.1002/ajh.23551. Epub 2013 Sep 12. PMID 23873804
- [Result] Bauchet L, Rigau V, Mathieu-Daude H, Figarella-Branger D, Hugues D, Palusseau L, Bauchet F, Fabbro M, Campello C, Capelle L, Durand A, Tretarre B, Frappaz D, Henin D, Menei P, Honnorat J, Segnarbieux F. French brain tumor data bank: methodology and first results on 10,000 cases. J Neurooncol. 2007 Sep;84(2):189-99. doi: 10.1007/s11060-007-9356-9. Epub 2007 Apr 13. PMID 17431547